CLINICAL TRIAL: NCT04508504
Title: Pericapsular Nerve Group (PENG) Block for Arthroscopic Hip Surgery: A Randomized, Placebo-controlled Trial
Brief Title: PENG Block for Arthroscopic Hip Surgery
Acronym: PENG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Peter Amato, MD, Assistant Professor of Anesthesiology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSR200214
Record Dates: First submitted 2020-07-25; First posted 2020-08-11 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Pain; Hip Arthroscopy
Keywords: pericapsular nerve group block, PENG, hip arthroscopy, pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized to one of two groups with a computer generated arm assignment. The sealed envelopes will be opened immediately prior to nerve block. One group will receive a PENG block and the other will receive a placebo block. The provider performing the block will not be blinded, however all other members of the care team, the patient, and the investigator collecting data will be blinded to the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preop PENG Block (Experimental): Patients will receive a preoperative ultrasound-guided pericapsular nerve group block with 20 mL 0.5% ropivacaine in a manner consistent with Girón-Arango et al 2018 (PMID:30063657). Using appropriate sterile precautions, and procedural sedation with up to 2 mg IV midazolam, an ultrasound (SonoSite S-Nerve or Export) equipped with either a linear 15-6 megahertz (MHz), or a curvilinear 5-2 MHz transducer (habitus-dependent) is used to identify the anterior inferior iliac spine, iliopubic eminence, and psoas muscle. After skin localization with 1-2 mL 1% lidocaine, a 22g 80 mm echogenic block needle (Pajunk SonoBlock II Facet) is advanced lateral to medial, in plane with the ultrasound beam, beneath the psoas tendon to the iliopubic eminence. 20 mL 0.5% ropivacaine is injected beneath the psoas tendon and above the iliopubic eminence, in 5 mL increments with periodic aspiration to prevent intravascular injection. The needle is withdrawn, and the needle entry site wiped clean.
  Interventions: Procedure: Preop PENG block; Drug: Ropivacaine 0.5% Injectable Solution
- Placebo (Placebo Comparator): Patients in the placebo group will receive a subcutaneous injection of 5 mL 0.9% normal saline. Using appropriate sterile precautions, and procedural sedation with up to 2 mg IV midazolam, an ultrasound (SonoSite S-Nerve or Export) equipped with either a linear 15-6 megahertz (MHz), or a curvilinear 5-2 MHz transducer (habitus-dependent) is used to identify the anterior inferior iliac spine, iliopubic eminence, and psoas muscle. After skin localization with 1-2 mL 1% lidocaine, a 22g 80 mm echogenic block needle (Pajunk SonoBlock II Facet) is advanced lateral to medial, in plane with the ultrasound beam, 1-2 cm beneath the skin, remaining in the subcutaneous tissue. 5 mL of 0.9% normal saline is injected, with periodic aspiration to prevent intravascular injection. The needle is withdrawn, and the needle entry site wiped clean.
  Interventions: Procedure: Placebo block; Drug: Normal Saline

INTERVENTIONS:
Procedure: Preop PENG block — Ultrasound-guided injection of 20 mL 0.5% ropivacaine according to the method described by Giron-Arango L in 2018. A needle is inserted at the inguinal level under ultrasound guidance to pass beneath the psoas tendon on top of the iliopubic eminence where the local anesthetic is injected.
  Other Names: Pericapsular nerve group block
  Arms: Preop PENG Block
Procedure: Placebo block — Ultrasound-guided placebo injection of 5 mL 0.9% normal saline. Using the same landmarks as for the PENG group, a needle is inserted in the inguinal region under ultrasound guidance, whereby a subcutaneous injection of 5 mL of 0.9% saline is made.
  Arms: Placebo
Drug: Ropivacaine 0.5% Injectable Solution — 20 mL 0.5% ropivacaine will be injected for the preop PENG block
  Arms: Preop PENG Block
Drug: Normal Saline — 5 mL 0.9% Normal saline will be injected for the Placebo block
  Arms: Placebo

SUMMARY:
This randomized, double-blinded, placebo-controlled trial seeks to evaluate the analgesic efficacy of the pericapsular nerve group block in the setting of outpatient hip arthroscopy.

DETAILED DESCRIPTION:
The pericapsular nerve group, or PENG block, has been recently described and shows promise in providing analgesia to the hip joint. The analgesic value of this block in the setting of hip arthroscopy is unknown. This study aims to compare a preoperative PENG block to placebo block prior to outpatient hip arthroscopy under general anesthesia. The primary outcome measure is immediate postoperative pain as measured by numerical rating score in the post-anesthesia care unit (PACU). Secondary outcomes include opioid consumption, opioid-related adverse events, patient satisfaction, chronic opioid usage, and pain scores at other time points.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old undergoing unilateral hip arthroscopy at the outpatient surgery center.

Exclusion Criteria:

* refusal to participate
* < 18 yo
* Chronic opioid use
* localized infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
PACU pain score | Within 30 minutes of emergence from anesthesia.
  Maximum pain score within the first 30 minutes after emergence in the post-anesthesia care unit. Pain will be assessed by numerical rating score (0-10, where 0 is no pain, and 10 is the worst possible pain).

SECONDARY OUTCOMES:
PACU opioid consumption | Beginning with emergence from anesthesia and ending with discharge from the post-anesthesia care unit (typically 2 hours).
  Total morphine milligram equivalents required by patients in the post-anesthesia care unit, prior to discharge from the outpatient surgery center. Following emergence from anesthesia, pain will be assessed in regular intervals, with administration of IV and oral opioids according to numeric rating scale and clinical assessment. Opioid administration stops when patient numerical rating score is <4, when patient endorses manageable pain level, when side effects of opioids are intolerable, or for other concerning clinical conditions as determined by the anesthesiologist of record.
Nausea and Vomiting | Beginning with emergence from anesthesia and ending with discharge from the post-anesthesia care unit (typically 2 hours).
  This is a yes/no binary outcome measure defined by administration of any antiemetic drug in the post-anesthesia care unit.
Patient satisfaction with analgesia | Determined through follow-up calls at 24 hours and 48-hours.
  Patients will be called at 24 hours and 48 hours postoperatively. They will be asked during each call if they are satisfied with their pain control (binary - yes or no).
Postoperative opioid utilization | Determined through follow-up calls at 24 hours, 48 hours, and 1 week postoperatively
  Cumulative postoperative opioid consumption expressed in morphine milligram equivalents
Postoperative pain scores | Determined through follow-up calls at 24 hours, 48 hours, and 1 week postoperatively
  Postoperative numerical rating scores after discharge (0-10, where 0 is no pain, and 10 is the worst possible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Peter E Amato, MD, Principal Investigator — University of Virginia
Locations (1):
- UVA Outpatient Surgery Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Derived] Amato PE, Coleman JR, Dobrzanski TP, Elmer DA, Gwathmey FW Jr, Slee AE, Hanson NA. Pericapsular nerve group (PENG) block for hip arthroscopy: a randomized, double-blinded, placebo-controlled trial. Reg Anesth Pain Med. 2022 Aug 23:rapm-2022-103907. doi: 10.1136/rapm-2022-103907. Online ahead of print. PMID 35998937

DOCUMENTS (1):
  • Informed Consent Form (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT04508504/ICF_000.pdf